CLINICAL TRIAL: NCT04201704
Title: Effect of Restricted Fluid Management Strategy on Outcomes in Critically Ill Pediatric Trauma Patients: A Multicenter Randomized Controlled Trial
Brief Title: Effect of Giving Reduced Fluid in Children After Trauma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Northwell Health (Other); Johns Hopkins University (Other); Cornell University (Other); Childress Institute for Pediatric Trauma (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAR2083
Record Dates: First submitted 2019-12-12; First posted 2019-12-17 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Critical Illness; Pediatrics; General Surgery; Fluid Therapy; Wounds and Injuries
Keywords: Fluid Therapy; Intensive Care Units, Pediatric; Critical Care; Wounds and Injuries; Multiple Trauma; Treatment Outcome; Postoperative Complications; Resuscitation; Hemodynamics; Infusions, Intravenous; Isotonic Solutions; Crystalloid Solutions; Diuretics; Organism Hydration Status; Body Water
MeSH Terms: conditions — Critical Illness; Wounds and Injuries; Multiple Trauma; Postoperative Complications | interventions — Ringer's Lactate; Plasma Volume

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liberal IV Fluid (Active Comparator): * Maintenance fluid rate calculated by 4-2-1 formula for patients <110kg: 4 mL/kg for first 0-10kg + 2 mL/kg for 11-20kg + 1 mL/kg for each kg >20kg
  * Patients >110kg maintenance 150 mL/hr
  * Bolus Criteria: change in 1 of: >20% decrease in systolic blood pressure 50th percentile for age and sex, >20% increase in heart rate over 50th percentile for age, base excess > -5mmol/L, blood lactate >2mmol/L, AND urine output (UO) <1 mL/kg/hr if <50kg or <50 mL/hr if >50kg
  * If criteria met: bolus 20 mL/kg if <50kg or 1 L if ≥50 kg
  * For transfusion: give 10 mL/kg packed red blood cells, platelets, or fresh frozen plasma up to 250 mL. If >25kg give 250 mL.
  * Diuresis- after minimum 24hrs: if UO <2 mL/kg/hr (or <100 mL/hr if >50 kg) continue maintenance rate and bolus per initial phase. If UO >2 mL/kg/hr (or >100 mL/hr if >50kg), and lactate, systolic blood pressure, heart rate, creatinine are normal then lower IV fluid rate to ½ maintenance rate and then to "keep vein open" once on regular feeds
  Interventions: Other: Balanced crystalloid solution volume administration; Other: Packed Erythrocytes Units, Blood Product Unit volume; Other: Plasma volume; Other: Platelets volume
- Restricted IV Fluid (Experimental): * Maintenance fluid rate calculated by 70% of 4-2-1 formula if <110 kg: 4 mL/kg for first 0-10 kg, + 2 mL/kg for 11-20 kg, + 1 mL/kg for every kg >20 kg
  * Patients >110 kg: maintenance is 105 mL/hr
  * If same bolus criteria met: 10 mL/kg for patients <50kg, or 500 mL if ≥50 kg
  * If meet transfusion criteria: transfuse 10 mL/kg with packed red blood cells, platelets, or fresh frozen plasma by weight up to 250 mL. Patients >25 kg get 250 mL per transfusion
  * Diuresis (after minimum 24 hrs): if UO <1 mL/kg/hr (or <50 mL/hr if >50 kg) then continue IV fluids at maintenance rate and bolus as needed. If UO 1-2 mL/kg/hr (or 50-100 mL/hr if >50 kg) then decrease IV rate to ½ maintenance rate. If UO >2 mL/kg/hr (or >100 mL/hr if >50 kg), and Lactate, systolic blood pressure, heart rate, creatinine normal then reduce to "keep vein open" and consider Furosemide for goal UO >2-4 mL/kg/hr (100-200 mL/hr if >50 kg) until euvolemic
  Interventions: Other: Balanced crystalloid solution volume administration; Other: Packed Erythrocytes Units, Blood Product Unit volume; Other: Plasma volume; Other: Platelets volume

INTERVENTIONS:
Other: Balanced crystalloid solution volume administration — Maintenance and bolus fluid volumes of balanced isotonic crystalloid solution administered based on arm.
  Other Names: lactated ringers
Other: Packed Erythrocytes Units, Blood Product Unit volume — For patients designated as Bleeding, where hemoglobin <7 then patient will be transfused 10 mL/kg up to 250 mL/transfusion. If patient is hypovolemic with clinician discretion transfuse 20 mL/kg.
Other: Plasma volume — For patients designated as Bleeding, where International Normalized Ratio (INR) > 1.5 then patient will be transfused 10 mL/kg up to 250 mL/transfusion. If patient is hypovolemic with clinician discretion transfuse 20 mL/kg.
Other: Platelets volume — For patients designated as Bleeding, where platelets < 50,000 then patient will be transfused 10 mL/kg up to 250 mL/transfusion. If patient is hypovolemic with clinician discretion transfuse 20 mL/kg.

SUMMARY:
This study is designed to help decide how much intravenous (IV) fluid should be given to pediatric trauma patients. No standard currently exists for managing fluids in critically ill pediatric trauma patients, and many fluid strategies are now in practice. For decades, trauma patients got high volumes of IV fluid. Recent studies in adults show that patients actually do better by giving less fluid. The investigators do not know if this is true in children and this study is designed to answer that question and provide guidelines for IV fluid management in children after trauma.

DETAILED DESCRIPTION:
Aggressive fluid resuscitation has been the cornerstone of early post-operative and trauma management for decades. However, recent prospective adult studies have challenged this practice, linking high volume crystalloid resuscitation to increased mortality, cardiopulmonary, gastrointestinal and hematologic complications. A retrospective study the investigators recently performed at their quaternary-care children's hospital echoed these results. High quality prospective data is necessary to determine best practice guidelines in our pediatric surgery and trauma patients.

Currently, no standard exists to guide management of crystalloid fluid administration in trauma patients. Both liberal and restricted strategies are in use, dependent on physician discretion. The investigators propose the first randomized controlled trial (RCT) comparing a liberal to a restricted fluid management strategy in critically ill pediatric trauma patients. The objective of this comparative effectiveness study is to conduct a multicenter (around 10 sites) randomized controlled trial (RCT) to determine whether liberal or restricted fluid administration leads to better outcomes in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Trauma patients older than 6 months and younger than 15 years admitted to the pediatric intensive care unit (PICU)
* Patients admitted to the PICU directly from the Emergency Department (ED)
* Patients admitted to the PICU from the operating room (OR)
* Patients transferred to PICU from outside facility ED (need to have been in ED 12 hours or less)

Exclusion Criteria:

* Patients transferred to PICU from outside PICU or inpatient floor
* Patients transferred to PICU from outside facility ED if >12 hours
* Patients expected to be discharged from the PICU within 24 hours
* Patient with congenital heart disease as defined by a congenital cardiac defect requiring surgery or medication
* Patient with diagnosis of chronic cardiac condition (e.g. hypertension, cardiac arrhythmia)
* Patients with chronic kidney disease as defined by an abnormality of kidney structure or function, present for more than 3 months, with implications to health
* Post-operative transplant, cardiac, and neurosurgical patients
* Patients with traumatic brain injury
* Patients with any disease that may affect baseline blood pressure and heart rate (endocrine disorders, certain genetic disorders, mitochondrial diseases)
* Hypotension requiring vasopressor therapy
* If massive transfusion protocol initiated

Ages: 6 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2018-08-27 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Overall complications | Up to time of discharge (up to approximately 1 month)
  Total number of complications defined as pulmonary edema, hemorrhage, deep cavity infection, anastomotic dehiscence, thrombosis, death, superficial wound infection, ileus, and pneumonia.

SECONDARY OUTCOMES:
Number of Hours of Hospital Length of Stay | Up to time of discharge (up to approximately 1 month)
  length of time in hospital to inpatient discharge in hours
Number of Hours of ICU Length of Stay | Up to time of discharge (up to approximately 1 month)
  length of time in pediatric intensive care unit in hours
Number of hours on Supplemental Oxygen | Up to time of discharge (up to approximately 1 month)
  length of time patient requires non-invasive supplemental O2 in hours
Number of Hours on Ventilator | Up to time of discharge (up to approximately 1 month)
  length of time patient requires invasive ventilation in hours

CONTACTS AND LOCATIONS:
Overall Officials: Vincent P Duron, MD, Principal Investigator — Columbia University
Locations (4):
- United States (4):
  - John R. Oishei Children's Hospital of Buffalo, Buffalo, New York
  - Columbia University Irving Medical Center NewYork-Presbyterian Morgan Stanley Children's Hospital, New York, New York
  - University of Rochester, Golisano Children's Hospital, Rochester, New York
  - Le Bonheur Children's Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bickell WH, Wall MJ Jr, Pepe PE, Martin RR, Ginger VF, Allen MK, Mattox KL. Immediate versus delayed fluid resuscitation for hypotensive patients with penetrating torso injuries. N Engl J Med. 1994 Oct 27;331(17):1105-9. doi: 10.1056/NEJM199410273311701. PMID 7935634
- [Background] Arikan AA, Zappitelli M, Goldstein SL, Naipaul A, Jefferson LS, Loftis LL. Fluid overload is associated with impaired oxygenation and morbidity in critically ill children. Pediatr Crit Care Med. 2012 May;13(3):253-8. doi: 10.1097/PCC.0b013e31822882a3. PMID 21760565
- [Background] Bouchard JE, Mehta RL. Fluid balance issues in the critically ill patient. Contrib Nephrol. 2010;164:69-78. doi: 10.1159/000313722. Epub 2010 Apr 20. PMID 20427995
- [Background] Coons BE, Tam S, Rubsam J, Stylianos S, Duron V. High volume crystalloid resuscitation adversely affects pediatric trauma patients. J Pediatr Surg. 2018 Nov;53(11):2202-2208. doi: 10.1016/j.jpedsurg.2018.07.009. Epub 2018 Jul 24. PMID 30072215
- [Background] Cotton BA, Guy JS, Morris JA Jr, Abumrad NN. The cellular, metabolic, and systemic consequences of aggressive fluid resuscitation strategies. Shock. 2006 Aug;26(2):115-21. doi: 10.1097/01.shk.0000209564.84822.f2. PMID 16878017
- [Background] Feinman M, Cotton BA, Haut ER. Optimal fluid resuscitation in trauma: type, timing, and total. Curr Opin Crit Care. 2014 Aug;20(4):366-72. doi: 10.1097/MCC.0000000000000104. PMID 24979715
- [Background] Fletcher JJ, Bergman K, Blostein PA, Kramer AH. Fluid balance, complications, and brain tissue oxygen tension monitoring following severe traumatic brain injury. Neurocrit Care. 2010 Aug;13(1):47-56. doi: 10.1007/s12028-010-9345-2. PMID 20376708
- [Background] Foland JA, Fortenberry JD, Warshaw BL, Pettignano R, Merritt RK, Heard ML, Rogers K, Reid C, Tanner AJ, Easley KA. Fluid overload before continuous hemofiltration and survival in critically ill children: a retrospective analysis. Crit Care Med. 2004 Aug;32(8):1771-6. doi: 10.1097/01.ccm.0000132897.52737.49. PMID 15286557
- [Background] Kasotakis G, Sideris A, Yang Y, de Moya M, Alam H, King DR, Tompkins R, Velmahos G; Inflammation and Host Response to Injury Investigators. Aggressive early crystalloid resuscitation adversely affects outcomes in adult blunt trauma patients: an analysis of the Glue Grant database. J Trauma Acute Care Surg. 2013 May;74(5):1215-21; discussion 1221-2. doi: 10.1097/TA.0b013e3182826e13. PMID 23609270
- [Background] Klein MB, Hayden D, Elson C, Nathens AB, Gamelli RL, Gibran NS, Herndon DN, Arnoldo B, Silver G, Schoenfeld D, Tompkins RG. The association between fluid administration and outcome following major burn: a multicenter study. Ann Surg. 2007 Apr;245(4):622-8. doi: 10.1097/01.sla.0000252572.50684.49. PMID 17414612
- [Background] Ley EJ, Clond MA, Srour MK, Barnajian M, Mirocha J, Margulies DR, Salim A. Emergency department crystalloid resuscitation of 1.5 L or more is associated with increased mortality in elderly and nonelderly trauma patients. J Trauma. 2011 Feb;70(2):398-400. doi: 10.1097/TA.0b013e318208f99b. PMID 21307740
- [Background] National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome (ARDS) Clinical Trials Network; Wiedemann HP, Wheeler AP, Bernard GR, Thompson BT, Hayden D, deBoisblanc B, Connors AF Jr, Hite RD, Harabin AL. Comparison of two fluid-management strategies in acute lung injury. N Engl J Med. 2006 Jun 15;354(24):2564-75. doi: 10.1056/NEJMoa062200. Epub 2006 May 21. PMID 16714767
- [Background] Owens TM, Watson WC, Prough DS, Uchida T, Kramer GC. Limiting initial resuscitation of uncontrolled hemorrhage reduces internal bleeding and subsequent volume requirements. J Trauma. 1995 Aug;39(2):200-7; discussion 208-9. doi: 10.1097/00005373-199508000-00004. PMID 7674386
- [Background] Takil A, Eti Z, Irmak P, Yilmaz Gogus F. Early postoperative respiratory acidosis after large intravascular volume infusion of lactated ringer's solution during major spine surgery. Anesth Analg. 2002 Aug;95(2):294-8, table of contents. doi: 10.1097/00000539-200208000-00006. PMID 12145036
- [Background] Watters JM, Tieu BH, Todd SR, Jackson T, Muller PJ, Malinoski D, Schreiber MA. Fluid resuscitation increases inflammatory gene transcription after traumatic injury. J Trauma. 2006 Aug;61(2):300-8; discussion 308-9. doi: 10.1097/01.ta.0000224211.36154.44. PMID 16917442
- [Background] Leteurtre S, Martinot A, Duhamel A, Proulx F, Grandbastien B, Cotting J, Gottesman R, Joffe A, Pfenninger J, Hubert P, Lacroix J, Leclerc F. Validation of the paediatric logistic organ dysfunction (PELOD) score: prospective, observational, multicentre study. Lancet. 2003 Jul 19;362(9379):192-7. doi: 10.1016/S0140-6736(03)13908-6. PMID 12885479
- [Derived] Duron VP, Ichinose R, Stewart LA, Porigow C, Fan W, Rubsam JM, Stylianos S, Dorrello NV. Pilot randomized controlled trial of restricted versus liberal crystalloid fluid management in pediatric post-operative and trauma patients. Pilot Feasibility Stud. 2023 Nov 8;9(1):185. doi: 10.1186/s40814-023-01408-w. PMID 37941073